CLINICAL TRIAL: NCT02502305
Title: Liveonline Training Course to Improve Food Habits and Enhance Physical Activity in Older Adults
Acronym: LIFE!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Liveonline Coaching (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Professor of Health Psychology, Jacobs University Bremen gGmbH
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUFP7-30583JUB
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Impaired Health; Motivation
Keywords: health literacy; attitude; motivation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): intervention group receives liveonline course training, 3 questionnaires at an interval of 6 weeks
  Interventions: Behavioral: liveonline course
- Control group (No Intervention): control group receives 3 questionnaires at an interval of 6 weeks

INTERVENTIONS:
Behavioral: liveonline course — physical activity and healthy diet are targeted and should be enhanced, health literacy (HL) in older people should be improved
  Arms: Intervention group

SUMMARY:
Aim of the study is to find out if the live online course is effective with regard to health promotion. Older adults receive support to initiate a health behavior (i.e., to enhance physical activity or to improve food habits).

Motivation, confidence and self-management strategies are optimized to make sure participants are able to integrate the physical activity or healthy diet into their daily life.

DETAILED DESCRIPTION:
Aim of the study is to support older adults to define a personal health behavior (to enhance physical activity, to improve food habits), to check and optimize this intention regarding self-efficacy and volitional competencies, such as action and coping planning, disability management to adopt and maintain their behavior successfully.

Research questions:

* What is the pathway from health information/intention to behavioural change (motivational and volitional processes)?
* Which are the crucial social-cognitive variables in educating/coaching adults with low health literacy in daily self-management?
* Which other resources (e.g. social support) should be targeted in interventions to empower people in health behaviour change and maintenance?

ELIGIBILITY:
Inclusion Criteria:

* internet access at home
* proficient language skills (German)

Exclusion Criteria:

* no internet access at home
* no proficient language skills (German)
* contra-indication for physical activity or a diet rich in fruit and vegetables

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
health literacy | up to 4 months
  health literacy will be assessed by questions in a questionnaire

SECONDARY OUTCOMES:
physical activity | up to 4 months
  physical activity will be assessed by questions in a questionnaire
healthy diet | up to 4 months
  healthy diet will be assessed by questions in a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Jacobs University Bremen gGmbH
Locations (1):
- Jacobs University Bremen gGmbH, Bremen, City state Bremen, Germany